CLINICAL TRIAL: NCT01356316
Title: Immunogenicity and Safety of a Trivalent Inactivated Influenza Vaccine, Formulation 2010-2011, in Non-Elderly Adult and Elderly Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Adimmune Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FLU10T11A
Record Dates: First submitted 2011-05-17; First posted 2011-05-19 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2012-12

CONDITIONS: Influenza
Keywords: Influenza; Vaccine; Immunogenicity
MeSH Terms: conditions — Influenza, Human

ARMS (1):
- AdimFlu-S Influenza Vaccine (Experimental)
  Interventions: Biological: AdimFlu-S Vaccine 2010-2011

INTERVENTIONS:
Biological: AdimFlu-S Vaccine 2010-2011 — Per ml contains following strains 30μg, A/California/7/2009 (H1N1), A/Perth/16/2009 (H3N2) and B/Brisbane/60/2008

SUMMARY:
Each potential subject will be screened before the start of the study to determine their eligibility for participation. Just prior to vaccination, a 10 mL venous blood sample will be taken from each eligible subject, for baseline titration of circulating anti-HA antibodies. Immediately thereafter, each subject received one dose of vaccine (0.5 mL) by intramuscular injection into the upper arm. Subjects will be asked to stay at the site for 30 minutes post-vaccination to observe for immediate reaction. Subjects will be monitored for adverse events during the study. At three weeks (±3 days) after the vaccination, subjects will be asked to return to the site for final collection of blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant females and aged ³ 18 years;
* Willing and able to adhere to visit schedules and all study requirements;
* Subjects read and signed the study-specific informed consent.

Exclusion Criteria:

* Subject or his/her family is employed by the participated hospital;
* Subjects received influenza vaccine (Trivalent and/or A(H1N1)) within the previous 6 months;
* History of hypersensitivity to eggs or egg protein or similar pharmacological effects to study medication;
* Personal or family history of Guillain-Barré Syndrome;
* An acute febrile illness within 1 week prior to vaccination;
* Current upper respiratory illness (URI), including the common cold or nasal congestion within 72 hours;
* Patients with influenza-like illness as defined by the presence of fever (temperature ≥38ºC) and at least two of the following four symptoms: headache, muscle/joint aches and pains (e.g. myalgia/arthralgia), sore throat and cough;
* Female subjects who are pregnant, lactating or likely to become pregnant during the study; Women of childbearing potential disagree to use an acceptable method of contraception (e.g., hormonal contraceptives, IUD, barrier device or abstinence) throughout the study.
* Treatment with an investigational drug or device, or participation in a clinical study, within 3 months before consent;
* Immunodeficiency, immunosuppressive or household contact with immunosuppression;
* History of wheezing or bronchodilator use within 3 months prior to study vaccine;
* Receipt of live virus vaccine within 1 month prior to study vaccine or expected receipt within 1 month of study vaccination;
* Receipt of any inactivated vaccine within 2 weeks prior to study vaccination or expected receipt within 1 month of study vaccination;
* Receipt of any blood products, including immunoglobulin in the prior 3 months;
* Underlying condition in the investigators' opinion may interfere with evaluation of the vaccine;
* Significant chronic illness for which inactivated influenza vaccine is recommended or commonly used.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-08; Primary Completion 2010-08 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The primary objective is to evaluate the immunogenicity profiles for influenza virus vaccine strains (2010-2011 season) of the AdimFlu-S manufactured by Adimmune Corporation. | Change from baseline for anti-hemaglutinin (HA) antibodies by hemagglutinaton inhibition (HAI) at 21 days post immunization
  Twenty-one days after vaccination, serum samples will be taken and tested for anti-hemaglutinin (HA) antibodies by hemagglutinaton inhibition (HAI), and assays will be performed at Adimmune Corporation designated central laboratory. Subjects will be considered to be seronegative if serum HAI titer<1:10. The seroconversion is defined as the post-vaccination serum at least 40 for whom had negative pre-vaccination or a fourfold or greater increase in HAI titers in subjects who had positive pre-vaccination serum.

SECONDARY OUTCOMES:
The secondary objective is to evaluate the safety and tolerability profiles including the presence or absence of the pre-specified reactogenicity events and other serious/non-serious adverse events of the AdimFlu-S manufactured by Adimmune Corporation. | 7 days after vaccination
  Reactogenicity events are pre-specified adverse events systematically recorded on diary cards(a grid of check boxes for each event and each day) during the immediate post-vaccination period by all participants. In general, reactogenicity events will be recorded for 7 days after vaccination. The selection of the events to be collected systematically is based on events expected to occur with wild-type influenza infection.
  In regard to the long term safety of the study vaccine, the significant and/or serious adverse event(s) will be recorded during the 6 months follow up after vaccination.